CLINICAL TRIAL: NCT05724706
Title: An Evaluation of Salivary Oxidant and Antioxidant Levels in Peri-implant Health and Disease
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other); Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Zeynep Seda Pekcetin-Bayav, Assistant Professor Doctor, Biruni University
Other Study IDs: Z PEKCETIN-BAYAV
Record Dates: First submitted 2021-03-22; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Peri-Implantitis; Bone Loss in Jaw; Dental Implant Failed; Dental Implant Failure Nos; Oxidative Stress
Keywords: oxidant; antioxidant; oxidative stress; Peri-implantitis; Marginal bone loss
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — unstimulated saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with peri-implantitis (PI): The PI group consisted of 23 patients (9M/14F) with ages ranging from 29 to 66 years (mean 51,91 ± 10,63). This group was selected based on the success criteria of Misch et al. 2008; patients with clinical findings such as bleeding and/or sweeping in their implants, pain or tenderness during function, and exudation in peri-implant tissues, with at least 1 implant with a pocket depth of more than 7 mm and radiographic bone loss of at least 4 mm or more around the implant were included.
- Patients with marginal bone loss (MBL): The MBL group consisted of 22 patients (14M /8F) aged between 27 and 67 years (mean 53,00 ± 8,92). This group was based on the success criteria defined by Misch et al. 2008; patients for whom, in the clinical examination of implants, there was no bleeding, non-sweeping, non-mobility, with no exudation history of peri-implant tissues, no pain or sensitivity when in function, and there was at least 1 implant with 2-4 mm radiographic bone loss around the implant were included.
- Patients with healthy peri-implant tissues (HI): The HI group consisted of 22 patients(7M/15F) with ages ranging from 29 to 62 years (mean 51,00 ± 8,45). This group was based on the success criteria defined by Misch et al. in 2008: Patients with no history of exudation in the periimplant tissues, no bleeding and suppuration during probing, no pain or sensitivity in function, no mobility, and at least 1 implant with a radiographic bone loss around the implant of less than 2 mm were included.
- Healthy control (HC): 21 individuals (8M/ 13F) whose ages ranged between 27 and 67 (mean 21.88 ± 11.21 years), who did not have any dental implants, and who were selected among the patient community were included the study as a healthy control group (HC).

SUMMARY:
Objectives: Inflammatory lesions develop in the tissues surrounding implants are referred to as peri-implant diseases. Oxidants, play a role in inflammatory lesions. The study aimed to determine oxidant and antioxidant levels in the saliva of patients with various levels of peri-implant diseases and the relationship between oxidative stress and peri-implant diseases.

Material and methods: Sixty-seven patients with at least one dental implant applied in our clinic were included in the study. The patients were divided into 3 groups; with peri-implantitis (PI), with marginal bone loss (MBL) and with healthy peri-implant (HI) tissues. Twenty-one individuals who didn't have any dental implants were included the study as a healthy control group (HC). For oxidant concentration, total oxidant status (TOS), advanced oxidation protein products (AOPP), and for antioxidant concentration, total antioxidant status (TAS), were investigated.

DETAILED DESCRIPTION:
INTRODUCTION

Inflammatory lesions that develop in the tissues surrounding implants are generally referred to as peri-implant diseases. Peri-implant disease has two subgroups; peri-implant mucositis, which is reversible inflammatory lesion limited to the surrounding mucosal tissues, and peri-impantitis which is characterized by bone destruction around the dental implants. Peri-implant disease develops as a result of a balance problem between bacterial loading and host response around an implant that has been correctly secured by osseointegration. Bacteria produce tissue destruction directly, via toxic products, and indirectly, by activating host defense systems; in other words, by inflammation. Various types of molecules are formed in inflammatory lesions; these include reactive species such as free radicals (FR) and reactive oxygen species (ROS). ROS are physiological formations that are the endogenous sources of the mitochondrial electron transport chain seen in every living organism. ROS occur as a natural product of normal oxygen metabolism, and play an important role in cell signals and hemostasis. ROS increase during inflammation; hence, oxidizing conditions increase and cell structures are damaged. This condition is known as oxidative stress (OS). OS depends on an increase in FR production and/or a decrease in the protective mechanism (antioxidant status), and OS is defined as a balance problem between oxidants and antioxidants in the body.

Many studies support the idea that OS plays an important role in the etiology and severity of periodontal diseases.

The etiology and the pathogenic mechanism are similar in the periodontitis and peri-implant diseases processes. However, those studies indicating the effect of OS on peri-implant tissues have used quite small groups or small numbers of biomarkers. The results obtained have been contradictory.

Therefore, this study aimed to determine oxidant and antioxidant levels in the saliva of patients with various levels of peri-implant diseases and the relationship between oxidative stress and peri-implant diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older;
* Being systemically healthy; ,
* Being non-smokers;
* For dental implant groups, at least 1 osseointegrated implant;
* Dental implant applied by at least a specialist-level physician;
* Dental implants having the same surface and the same design;
* Correct prosthetic restoration of occlusal loading;
* Dental implant having been in function for at least 6 months.

Exclusion Criteria:

* Any history of medical conditions;
* Presence of active periodontal disease;
* Use of antibiotic or anti-inflammatory medications in the past 3 months;
* Pregnancy;
* Use of AO supplements;
* Smoking;
* Poor oral hygiene;
* Inflammation in the oral area;
* Presence of active caries;
* Presence of oral mucosal lesions such as oral lichen planus or recurrent aphthous stomatitis.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with peri-implantitis (PI); The PI group consisted of 23 patients (9M/14F) with ages ranging from 29 to 66 years
  Group 2: Patients with marginal bone loss (MBL); The MBL group consisted of 22 patients (14M /8F) aged between 27 and 67 years
  Group 3: Patients with healthy peri-implant tissues (HI); The HI group consisted of 22 patients(7M/15F) with ages ranging from 29 to 62 years
  Group 4: Healthy control (HC) 21 individuals (8M/ 13F) whose ages ranged between 27 and 67 years
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Identifying patients to be included in the study and collecting saliva samples | 1 year
  Patients to be included in the study were determined by clinical and radiological examinations, divided into groups, and saliva samples; it was collected to measure the total oxidant status (TOS) and advanced oxidation protein products (AOPP) to evaluate the oxidant concentration in it, and the total antioxidant status (TAS) to evaluate the antioxidant concentration in it and stored at -80 degrees Celsius.

SECONDARY OUTCOMES:
Biochemical examination of oxidant and antioxidant biomarkers in saliva and statistical evaluation of the results | 4 month
  In biochemical analysis, For oxidant concentration in saliva, total oxidant status (TOS), advanced oxidation protein products (AOPP), and for antioxidant concentration, total antioxidant status (TAS), were investigated. The values of markers whose biochemical analysis were made in saliva were statistically analyzed and calculated.
  Saliva TOS levels were reported as µM H2O2 equivalent per liter (µmol H2O2 Equiv/L).
  Saliva AOPP levels were reported as nmol / mL chloramine-T equivalent. Saliva TAS levels were reported as units of mM trolox equivalent per liter (mmol trolox Equiv/L).

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP S PEKCETIN-BAYAV, ASST. PROF., Study Director — Biruni University

IPD SHARING:
Plan to Share IPD: Undecided
It will be available when needed.

REFERENCES:
- [Background] Berglundh T, Persson L, Klinge B. A systematic review of the incidence of biological and technical complications in implant dentistry reported in prospective longitudinal studies of at least 5 years. J Clin Periodontol. 2002;29 Suppl 3:197-212; discussion 232-3. doi: 10.1034/j.1600-051x.29.s3.12.x. PMID 12787220
- [Background] Canakci CF, Cicek Y, Canakci V. Reactive oxygen species and human inflammatory periodontal diseases. Biochemistry (Mosc). 2005 Jun;70(6):619-28. doi: 10.1007/s10541-005-0161-9. PMID 16038603
- [Background] Chapple IL. Role of free radicals and antioxidants in the pathogenesis of the inflammatory periodontal diseases. Clin Mol Pathol. 1996 Oct;49(5):M247-55. doi: 10.1136/mp.49.5.m247. No abstract available. PMID 16696085
- [Background] Chapple IL. Reactive oxygen species and antioxidants in inflammatory diseases. J Clin Periodontol. 1997 May;24(5):287-96. doi: 10.1111/j.1600-051x.1997.tb00760.x. PMID 9178107
- [Background] Chapple IL, Brock G, Eftimiadi C, Matthews JB. Glutathione in gingival crevicular fluid and its relation to local antioxidant capacity in periodontal health and disease. Mol Pathol. 2002 Dec;55(6):367-73. doi: 10.1136/mp.55.6.367. PMID 12456773
- [Background] Chapple IL, Brock GR, Milward MR, Ling N, Matthews JB. Compromised GCF total antioxidant capacity in periodontitis: cause or effect? J Clin Periodontol. 2007 Feb;34(2):103-10. doi: 10.1111/j.1600-051X.2006.01029.x. Epub 2006 Dec 13. PMID 17214737
- [Background] Chapple IL, Matthews JB. The role of reactive oxygen and antioxidant species in periodontal tissue destruction. Periodontol 2000. 2007;43:160-232. doi: 10.1111/j.1600-0757.2006.00178.x. No abstract available. PMID 17214840
- [Background] Chapple IL, Milward MR, Ling-Mountford N, Weston P, Carter K, Askey K, Dallal GE, De Spirt S, Sies H, Patel D, Matthews JB. Adjunctive daily supplementation with encapsulated fruit, vegetable and berry juice powder concentrates and clinical periodontal outcomes: a double-blind RCT. J Clin Periodontol. 2012 Jan;39(1):62-72. doi: 10.1111/j.1600-051X.2011.01793.x. Epub 2011 Oct 17. PMID 22093005
- [Background] Chen AF, Chen DD, Daiber A, Faraci FM, Li H, Rembold CM, Laher I. Free radical biology of the cardiovascular system. Clin Sci (Lond). 2012 Jul;123(2):73-91. doi: 10.1042/CS20110562. PMID 22455351
- [Background] Edgar WM. Saliva: its secretion, composition and functions. Br Dent J. 1992 Apr 25;172(8):305-12. doi: 10.1038/sj.bdj.4807861. PMID 1591115
- [Background] Erel O. A novel automated direct measurement method for total antioxidant capacity using a new generation, more stable ABTS radical cation. Clin Biochem. 2004 Apr;37(4):277-85. doi: 10.1016/j.clinbiochem.2003.11.015. PMID 15003729
- [Background] Erel O. A new automated colorimetric method for measuring total oxidant status. Clin Biochem. 2005 Dec;38(12):1103-11. doi: 10.1016/j.clinbiochem.2005.08.008. Epub 2005 Oct 7. PMID 16214125
- [Background] Guo M, Liu L, Zhang J, Liu M. Role of Reactive Oxygen Species and Advanced Glycation End Products in the Malfunctioning of Dental Implants. West Indian Med J. 2015 Sep;64(4):419-23. doi: 10.7727/wimj.2014.105. Epub 2015 Apr 29. PMID 26624598
- [Background] Guncu GN, Tozum TF, Guncu MB, Yamalik N, Tumer C, Karabulut E, Kilinc K. Myeloperoxidase as a measure of polymorphonuclear leukocyte response in inflammatory status around immediately and delayed loaded dental implants: a randomized controlled clinical trial. Clin Implant Dent Relat Res. 2008 Mar;10(1):30-9. doi: 10.1111/j.1708-8208.2007.00058.x. PMID 18335584
- [Background] Hanasand M, Omdal R, Norheim KB, Goransson LG, Brede C, Jonsson G. Improved detection of advanced oxidation protein products in plasma. Clin Chim Acta. 2012 May 18;413(9-10):901-6. doi: 10.1016/j.cca.2012.01.038. Epub 2012 Feb 8. PMID 22336637
- [Background] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Background] Liskmann S, Vihalemm T, Salum O, Zilmer K, Fischer K, Zilmer M. Characterization of the antioxidant profile of human saliva in peri-implant health and disease. Clin Oral Implants Res. 2007 Feb;18(1):27-33. doi: 10.1111/j.1600-0501.2006.01296.x. PMID 17224020
- [Background] Liskmann S, Zilmer M, Vihalemm T, Salum O, Fischer K. Correlation of peri-implant health and myeloperoxidase levels: a cross-sectional clinical study. Clin Oral Implants Res. 2004 Oct;15(5):546-52. doi: 10.1111/j.1600-0501.2004.01061.x. PMID 15355396
- [Background] Liu Z, Liu Y, Song Y, Zhang X, Wang S, Wang Z. Systemic oxidative stress biomarkers in chronic periodontitis: a meta-analysis. Dis Markers. 2014;2014:931083. doi: 10.1155/2014/931083. Epub 2014 Nov 16. PMID 25477703
- [Background] Mehta M, Basalingappa K, Griffith JN, Andrade D, Babu A, Amreddy N, Muralidharan R, Gorospe M, Herman T, Ding WQ, Ramesh R, Munshi A. HuR silencing elicits oxidative stress and DNA damage and sensitizes human triple-negative breast cancer cells to radiotherapy. Oncotarget. 2016 Oct 4;7(40):64820-64835. doi: 10.18632/oncotarget.11706. PMID 27588488
- [Background] Misch CE. Contemporary Implant Dentistry. 3 rd ed. St. Louis, Missouri, Mosby; 2008.
- [Background] Mousavi Jazi M, Sadeghi Pour Rodsari HR, Mirmiran F. Level of Oxidative Stress Markers in Peri-Implant Crevicular Fluid and Their Correlation with Clinical Parameters. J Dent (Tehran). 2015 May;12(5):340-6. PMID 26877729
- [Background] Nagler RM, Klein I, Zarzhevsky N, Drigues N, Reznick AZ. Characterization of the differentiated antioxidant profile of human saliva. Free Radic Biol Med. 2002 Feb 1;32(3):268-77. doi: 10.1016/s0891-5849(01)00806-1. PMID 11827752
- [Background] Sanchez-Siles M, Lucas-Azorin J, Salazar-Sanchez N, Carbonell-Meseguer L, Camacho-Alonso F. Salivary Concentration of Oxidative Stress Biomarkers in a Group of Patients with Peri-Implantitis: A Transversal Study. Clin Implant Dent Relat Res. 2016 Oct;18(5):1015-1022. doi: 10.1111/cid.12367. Epub 2015 Jul 31. PMID 26230313
- [Background] Tonetti MS, Schmid J. Pathogenesis of implant failures. Periodontol 2000. 1994 Feb;4:127-38. doi: 10.1111/j.1600-0757.1994.tb00013.x. No abstract available. PMID 9673201
- [Background] Tunez I, Feijoo M, Huerta G, Montilla P, Munoz E, Ruiz A, Collantes E. The effect of infliximab on oxidative stress in chronic inflammatory joint disease. Curr Med Res Opin. 2007 Jun;23(6):1259-67. doi: 10.1185/030079907X187955. Epub 2007 Apr 25. PMID 17559725
- [Background] Zitzmann NU, Berglundh T. Definition and prevalence of peri-implant diseases. J Clin Periodontol. 2008 Sep;35(8 Suppl):286-91. doi: 10.1111/j.1600-051X.2008.01274.x. PMID 18724856
- [Background] Pietropaoli D, Ortu E, Severino M, Ciarrocchi I, Gatto R, Monaco A. Glycation and oxidative stress in the failure of dental implants: a case series. BMC Res Notes. 2013 Jul 26;6:296. doi: 10.1186/1756-0500-6-296. PMID 23890159